CLINICAL TRIAL: NCT00962910
Title: The European Quality of Care Pathways Study: The Impact of a Care Pathway for Proximal Femur Fracture (PFF) : an International Cluster Randomized Controlled Trial." (Www.E-P-A.Org)
Brief Title: European Quality of Care Pathways Study on Proximal Femur Fracture (EQCP-PFF)
Acronym: EQCP-PFF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: European Pathway Association (Other)
Collaborators: KU Leuven (Other); University of Eastern Piedmont (Other)
Responsible Party: Principal Investigator, Dr. Kris Vanhaecht, Dr. Kris Vanhaecht, Secretary General, European Pathway Association, ivzw, European Pathway Association
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: EPA-EQCP002
Record Dates: First submitted 2009-08-19; First posted 2009-08-20 (Estimated); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Femoral Fractures
Keywords: Femoral Fractures; Critical Pathway; Cluster Randomized Controlled Trial; Safety; Efficiency
MeSH Terms: conditions — Femoral Fractures | interventions — Critical Pathways

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pathway (Experimental): A care pathway will be implemented in this experimental group.
  Interventions: Other: PFF evidence based pathway
- Usual Care (No Intervention): Usual Care will be provided.

INTERVENTIONS:
Other: PFF evidence based pathway — A care pathway, as complex intervention, will be implemented.
  Other Names: pathway; care pathway; clinical pathway; critical pathway; integrated care pathway
  Arms: Pathway

SUMMARY:
Care pathways, a complex intervention to (re)organise, standardize and evaluate care processes, are used worldwide and in different kinds of settings. Although their international use, the impact is unclear. The European Quality of Care Pathways Study is the first international cluster Randomized Controlled Trial on the effect of care pathways for proximal femur fracture patients (PFF).

The hypothesis is that teams who work with care pathways for PFF patients deliver care that is more compliant to evidence based key interventions, have better patient outcomes and higher scores on team indicators than teams who do not work with care pathways.

DETAILED DESCRIPTION:
Healthcare is changing towards more patient focused care. The organization of the care process related to quality, efficiency and accessibility is one of the main areas of interest within the next years for clinicians, healthcare managers and policy makers. A main method to (re)organize a care process is the development and implementation of a care pathway. Care pathways, also known as clinical pathways or critical pathways, are used worldwide for a variety of patient groups. The European Pathway Association (E-P-A) defines a care pathway as: "A complex intervention for the mutual decision making and organization of predictable care for a well-defined group of patients during a well defined period. Defining characteristics of pathways includes: an explicit statement of the goals and key elements of care based on evidence, best practice and patient expectations; the facilitations of the communication and coordination of roles, and sequencing the activities of the multidisciplinary care team, patients and their relatives; the documentation, monitoring, and evaluation of variances and outcomes; and the identification of relevant resources".

Some prospective studies have been performed and published on the impact of pathways on quality and efficiency of care. The European Quality of Care Pathways (EQCP)-study will involve proximal femur fracture (PFF) to evaluate pathway effectiveness. Literature shows that adherence to international guidelines with regard to inhospital management of PFF is low for both pre-operative and post-operative care. Currently, some non-randomized trials (controlled clinical trials, cohort and case-control studies) and protocols about the impact of a care pathway for inpatient management of proximal femur fracture are published. The studies are conducted between 1992 and 2004, and the methodology is often doubtful. However, the studies indicate that care pathways for PFF improves performance with regard to pre-operative and post-operative interventions (i.e. time before surgery and time before mobilisation after surgery), and that they diminish length of stay (acute and total), in-hospital mortality, 30-day mortality, 1-year mortality, readmission rate and some post-operative complications like pressure sores or ulcers.

In the context of the high volume of PFF patients, high costs and high risk, and the complex coordination of care among multiple caregivers, a care pathway could enhance the quality of care in these patients by improving patient outcomes, promoting patient safety, increasing patient satisfaction, improving multidisciplinary teamwork and optimizing the use of resources.

The goal of the European Quality of Care Pathways (EQCP) study is:

* To evaluate the care pathway effectiveness in acute hospitals and their immediate link with primary care;
* To evaluate the effect of care pathways on team processes and team perceived organization of care.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria on cluster level are:

  1. Written agreement to participate in the study;
  2. Agreement that a care pathway for PFF will not be developed and used within the time frame of the study when randomized in the control group.
* Inclusion criteria on patient level are:

  1. Written informed consent;
  2. All consecutive admissions with PFF;
  3. Minimum age of 65 years;
  4. Closed fracture;
  5. Eligible for surgical intervention;
  6. ASA-score of 1, 2 or 3;
  7. Each patient was included only once in the study at initial hospitalization, even if the patient has been hospitalized more than once.

Exclusion Criteria:

* Exclusion criteria on patient level:

  1. Patients with severe dementia (DSM IV);
  2. Bone metastatic diseases (pathologic fractures);
  3. Second fracture on the same hip (i.e. peri-prosthetic fracture)

Inclusion criteria on multidisciplinary team level:

1. Team members are involved in direct patient care responsibilities for PFF;
2. Minimum representation of the core disciplines according to PFF literature;

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 514 (Actual)
Dates: Start 2009-05; Primary Completion 2014-05 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Mortality | 6 month

SECONDARY OUTCOMES:
Length of stay | in hospital
Pain score | in hospital

CONTACTS AND LOCATIONS:
Overall Officials: Kris Vanhaecht, PhD, Study Director — KU Leuven; Walter Sermeus, PhD, Principal Investigator — KU Leuven; Massimiliano Panella, PhD, Principal Investigator — Amedeo Avogadro University of Eastern Piemont

REFERENCES:
- [Derived] Handoll HH, Cameron ID, Mak JC, Panagoda CE, Finnegan TP. Multidisciplinary rehabilitation for older people with hip fractures. Cochrane Database Syst Rev. 2021 Nov 12;11(11):CD007125. doi: 10.1002/14651858.CD007125.pub3. PMID 34766330
- [Derived] Panella M, Seys D, Sermeus W, Bruyneel L, Lodewijckx C, Deneckere S, Sermon A, Nijs S, Boto P, Vanhaecht K. Minimal impact of a care pathway for geriatric hip fracture patients. Injury. 2018 Aug;49(8):1581-1586. doi: 10.1016/j.injury.2018.06.005. Epub 2018 Jun 4. PMID 29884319
- [Derived] Vanhaecht K, Sermeus W, Peers J, Lodewijckx C, Deneckere S, Leigheb F, Boonen S, Sermon A, Boto P, Mendes RV, Panella M; EQCP study group. The impact of care pathways for patients with proximal femur fracture: rationale and design of a cluster-randomized controlled trial. BMC Health Serv Res. 2012 May 24;12:124. doi: 10.1186/1472-6963-12-124. PMID 22640531
- See also: European Pathway Association — http://www.E-P-A.org